CLINICAL TRIAL: NCT06810180
Title: Examination of the Dynamic Relationships of Sleep, Physical Activity, and Circadian Rhythmicity With Neurobehavioral Heterogeneity in ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Keri Rosch, Clinical Psychologist/Associate Professor, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00478295
Record Dates: First submitted 2024-12-09; First posted 2025-02-05 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD); Sleep; Physical Activity
Keywords: ADHD; Circadian Rhythms; Ecological Momentary Assessment (EMA)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group (Experimental)
  Interventions: Behavioral: Go/No-Go Task; Behavioral: Delay discounting task; Behavioral: Mirror Tracing Persistence Task; Behavioral: Spatial Span; Behavioral: Stop Signal Task; Behavioral: Flanker task

INTERVENTIONS:
Behavioral: Go/No-Go Task — A computerized test in which participants are presented with red and green spaceship stimuli. They are told to press the spacebar in response to green spaceships (80% of trials) and withhold their response to red spaceships (20% of trials).
Behavioral: Delay discounting task — Participants make decisions between smaller, immediate rewards and larger, delayed rewards. The amount of the immediate reward and delay time are manipulated to identify individual delay discounting curves, or how the reward value decreases as a function of delay.
Behavioral: Mirror Tracing Persistence Task — A computerized test in which participants trace a star line drawing with a computer cursor using a trackpad with reversed directional controls. There are increasing levels of difficulty with participants being told they could quit the task during the very hard third star that they try to trace.
Behavioral: Spatial Span — Participants are instructed to attend to a computer screen to keep track of the order in which a happy face stimuli appears in a sequence of boxes positioned on the screen. They are presented with 2 trials at each level of difficulty, increasing from 2 stimuli by 1 additional stimuli per trial until they respond incorrectly for both trials within a level. There are two task conditions, forward and backward span, with the participant responding in the reverse order that the stimuli were presented for backward span.
Behavioral: Stop Signal Task — A computerized test in which participants are presented with a right or left facing arrow and are instructed to press a response button indicating the direction of the arrow. On 25% of the trials, an auditory beep is presented (i.e., stop signal) following the onset of the arrow (i.e., go signal) and participants are instructed to withhold their response when they hear the stop signal.
Behavioral: Flanker task — A computerized test in which a group of arrows are presented on the screen with the central arrow (target) pointing in the same/opposite direction as the 4 surrounding arrows (flankers). Participants are instructed to respond as quickly and accurately as possible to the central target arrow.

SUMMARY:
Attention deficit/hyperactivity disorder (ADHD) can present differently in individuals, with some individuals having difficulty with attentional control, hyperactivity, impulsivity, emotion dysregulation, and/or neurobehavioral functioning. The factors contributing to these different presentations remain unclear, but altered patterns of physical activity, sleep, and circadian rest/activity rhythms may play a key role.

The goal of this study is to leverage wearable technology (i.e., a wristband) to investigate the relationships between physical activity during the day, sleep patterns and disturbances, and 24-hour circadian rest/activity rhythms with differences in ADHD symptoms, emotion dysregulation, and related brain and behavioral features of attention-deficit/hyperactivity disorder (ADHD). The investigators hope this study will help improve assessment and intervention for individuals with ADHD by understanding how these factors relate to ADHD symptom expression and associated brain differences in ADHD.

Participants taking stimulant medication must withhold stimulant medication 24 hours before their research appointment and the morning of their research appointment. Stimulant medication may be restarted after the appointment is complete.

Participation in this study will require children to complete an initial 2-hour research appointment, two (2) weeks of activity and sleep monitoring at home using a wearable wristband and answering questions sent to a smartphone, and a second 4-hour research appointment after the 2-week period.

During the first research appointment, children will complete a cognitive assessment and a practice magnetic resonance imaging (MRI) scan. Parents/legal guardians will participate in the 30-45-minute sleep device training session with one of the research staff.

During the two weeks of activity/sleep monitoring at home, parents and children will answer questions about their sleep routine, ADHD symptoms, and emotional responding each morning and evening. Parents will be asked to install a questionnaire application on their smartphone. A prompt will be sent to their smartphone multiple times per day reminding parents to complete the brief assessment.

After the 2-week period, children will complete a 4-hour research appointment. During this research appointment, children will complete a 60-minute MRI scan and computer-based activities that assess cognitive skills, reward-based decision-making, and frustration tolerance. At the end of the research appointment, children will return the device to our research team. Parents may delete the questionnaire application from their phone at the end of the research appointment.

Participation will also require parents/legal guardians to complete questionnaires about their child. Questionnaires will be provided to the primary caregiver by email or at the beginning of their child's first research appointment. Parents agree to complete and return the questionnaires within one month of their child's research appointment.

Parents may be provided with additional questionnaires to give to their child's primary schoolteacher. This information is collected to better understand children's abilities, behavior, strengths, and weaknesses.

There are minimal risks associated with this study. Risks include fatigue, boredom, and mild discomfort.

There is no cost to participating in this study.

There is no direct benefit to participants for participating in this study.

ELIGIBILITY:
ADHD Clinical Group. Meet criteria for attention deficit/hyperactivity disorder (ADHD) according to DSM-5 criteria.

Exclusion Criteria:

Prematurity Prenatal exposure to alcohol or other substances Traumatic brain injury Co-occurring neurodevelopmental disorders (e.g., autism spectrum disorder, intellectual disability) Anxiety/mood disorders Active psychosis Bipolar disorder Conduct disorder Currently taking longer acting psychotropic medications that cannot be discontinued the day before research appointments

Control Group. Does not meet criteria for psychological or neuropsychological disorders Does not meet criteria for intellectual disability Does not meet criteria for a learning disorder

Exclusion Criteria:

Prematurity Prenatal exposure to alcohol or other substances Traumatic brain injury Currently taking medications that cannot be discontinued the day before research appointments

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Total Activity Counts (TAC) | Two-week, real-time period of at-home activity monitoring
  Using an actigraph, this study will collect daily physical activity levels of children. The actigraphic measure, total activity counts (TAC), will capture the number of times a child engages in periods of physical activity during the day and night.
Children's Sleep Health Questionnaire (CSHQ) Total Score | Within six months prior to the first research appointment.
  Sleep quality will be measured using the total score from the parent reported questionnaire asking about sleep duration, sleep disturbances, and sleep quality.
ADHD-related Symptoms | Within six months prior to the first research appointment.
  Parents will complete a diagnostic interview and rating scales reporting on ADHD symptoms, cognitive disengagement syndrome, irritability and emotion dysregulation.
Mean Fractional Anisotropy (FA) | Completed during the MRI scan on Day 15
  Mean fractional anisotropy (FA) is a structural connectivity diffusion weighted imaging outcomes. It is a value that represents the overall degree of directional diffusion within that area, with higher values indicating more organized/connectivity, aligned white matter fibers, and lower values suggesting less organized fibers.
  Mean fractional anisotropy (FA) will be assessed in six fronto-subcortical tracts of interest including (1) OFC-limbic striatum, (2) dlPFC-executive striatum, (3) ACC-limbic striatum, (4) ACC-executive striatum, (5) OFC- and (6) ACC-amygdala in each hemisphere.
Stop Signal Reaction Time | Task will be completed on Day 15
  Measure of inhibitory control from the stop signal task based on the mean stop signal delay and mean go reaction time.
Congruency Effect on Reaction Time | Task will be completed on Day 15
  Difference in reaction time on correct response trials from the flanker task with congruent versus incongruent flanking stimuli.
Commission Errors | Task will be completed on Day 15
  Percentage of incorrect responses on no-go trials during the go/no-go task.
Backward Span Accuracy | Task will be completed on Day 15
  Total number of correct trials for the digit and spatial span tasks (separately), backwards span condition
Delay Discounting Area Over the Curve (AOC) | Task will be completed on Day 15
  Area over the curve (AOC) is a measure of the extent to which an individual discounts a reward as a function of delay. We will assess this measure during delay discounting tasks with different types of rewards (money and game time).
Mirror Tracing Persistance Task Latency to Quit | Task will be completed on Day 15
  During the very hard star condition of the MTPT, participants may choose to quit the task. This is the amount of time that passes until they quit the task.
Total Sleep Time (TST) | Two-week, real-time period of at-home activity monitoring
  Total sleep time (TST) will be collected using a wearable actigraph wristband. This variable is reported in minutes.
Wake After Sleep Onset (WASO) | Two-week, real-time period of at-home activity monitoring
  This variable is collected using a wearable actigraph wristband. This variable is reported in minutes.
Sleep Efficiency | Two-week, real-time period of at-home activity monitoring
  This variable is collected using a wearable actigraph wristband. This variable is the proportion of time-in-bed spent asleep compared to the total time spent in bed.
Sleep Onset Latency (SOL) | Two-week, real-time period of at-home activity monitoring
  This variable is collected using a wearable actigraph wristband. This variable captures how long it takes for a child to fall asleep once they are in bed.
Intra-daily Variability | Two-week, real-time period of at-home activity monitoring
  This variable is collected using a wearable actigraph wristband. Intra-daily variability is a measure of how fragmented a person's rest-activity rhythm (RAR) is over the course of a 24-hour period. quantifies the amount of switching between high and low activity levels within a day. Higher IV values indicate greater fragmentation, which can be a sign of frequent napping or inefficient sleep.
Midline Estimating Statistic of Rhythm (MESOR) | Two-week, real-time period of at-home activity monitoring
  This variable is collected using a wearable actigraph wristband. Mesor is a rhythm-adjusted mean that describes the value around which a fitted wave oscillates. The wave is dictated by the intensity of physical activity over a 24-hour period.
Functional connectivity Z-scores | Completed during an MRI scan on Day 15
  Functional connectivity will be examined among the same 6 fronto-subcortical tracts of interest including (1) OFC-limbic striatum, (2) dlPFC-executive striatum, (3) ACC-limbic striatum, (4) ACC-executive striatum, (5) OFC- and (6) ACC-amygdala in each hemisphere, as well as within- and between-network connectivity of the default mode network with the frontoparietal, salience, and affective networks. The primary measure of functional connectivity will be derived by correlating the average time series across ROIs and converting the correlations to z scores using Fisher's transform.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hugo W. Moser Research Institute at Kennedy Krieger, Baltimore, Maryland
  - Kennedy Krieger Institute, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data collected through questionnaires, computer-tasks, and neuroimaging will be shared with the NIH National Data Archive in compliance with the current data sharing policies. De-identified participant-level data may include the summary metrics produced or extracted from the instruments used in this study.
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be available every six months from the date of initial recruitment through the requisite data sharing period specified in the grant terms. Data will be hosted by the NIH National Data Archive using the existing data structures, making it accessible to the scientific community.
Access Criteria: Data will be hosted by the NIH National Data Archive using the existing data structures, making it accessible to researchers who have an account and verified institutional affiliation. The de-identified IPD will be available throughout the duration of the study and for any requisite time after the conclusion of the study, as per NIH policy.
  Researchers interested in accessing the IPD can use the NIH NDA data package tool to select and download the summary data of interest.
  Identifiable data will not be available for sharing.

REFERENCES:
- [Background] Sibley MH, Arnold LE, Swanson JM, Hechtman LT, Kennedy TM, Owens E, Molina BSG, Jensen PS, Hinshaw SP, Roy A, Chronis-Tuscano A, Newcorn JH, Rohde LA; MTA Cooperative Group. Variable Patterns of Remission From ADHD in the Multimodal Treatment Study of ADHD. Am J Psychiatry. 2022 Feb;179(2):142-151. doi: 10.1176/appi.ajp.2021.21010032. Epub 2021 Aug 13. PMID 34384227
- [Background] Mordre M, Groholt B, Kjelsberg E, Sandstad B, Myhre AM. The impact of ADHD and conduct disorder in childhood on adult delinquency: a 30 years follow-up study using official crime records. BMC Psychiatry. 2011 Apr 11;11:57. doi: 10.1186/1471-244X-11-57. PMID 21481227
- [Background] Fredriksen M, Dahl AA, Martinsen EW, Klungsoyr O, Faraone SV, Peleikis DE. Childhood and persistent ADHD symptoms associated with educational failure and long-term occupational disability in adult ADHD. Atten Defic Hyperact Disord. 2014 Jun;6(2):87-99. doi: 10.1007/s12402-014-0126-1. Epub 2014 Feb 5. PMID 24497125
- [Background] Faraone SV, Banaschewski T, Coghill D, Zheng Y, Biederman J, Bellgrove MA, Newcorn JH, Gignac M, Al Saud NM, Manor I, Rohde LA, Yang L, Cortese S, Almagor D, Stein MA, Albatti TH, Aljoudi HF, Alqahtani MMJ, Asherson P, Atwoli L, Bolte S, Buitelaar JK, Crunelle CL, Daley D, Dalsgaard S, Dopfner M, Espinet S, Fitzgerald M, Franke B, Gerlach M, Haavik J, Hartman CA, Hartung CM, Hinshaw SP, Hoekstra PJ, Hollis C, Kollins SH, Sandra Kooij JJ, Kuntsi J, Larsson H, Li T, Liu J, Merzon E, Mattingly G, Mattos P, McCarthy S, Mikami AY, Molina BSG, Nigg JT, Purper-Ouakil D, Omigbodun OO, Polanczyk GV, Pollak Y, Poulton AS, Rajkumar RP, Reding A, Reif A, Rubia K, Rucklidge J, Romanos M, Ramos-Quiroga JA, Schellekens A, Scheres A, Schoeman R, Schweitzer JB, Shah H, Solanto MV, Sonuga-Barke E, Soutullo C, Steinhausen HC, Swanson JM, Thapar A, Tripp G, van de Glind G, van den Brink W, Van der Oord S, Venter A, Vitiello B, Walitza S, Wang Y. The World Federation of ADHD International Consensus Statement: 208 Evidence-based conclusions about the disorder. Neurosci Biobehav Rev. 2021 Sep;128:789-818. doi: 10.1016/j.neubiorev.2021.01.022. Epub 2021 Feb 4. PMID 33549739
- [Background] Hvolby A. Associations of sleep disturbance with ADHD: implications for treatment. Atten Defic Hyperact Disord. 2015 Mar;7(1):1-18. doi: 10.1007/s12402-014-0151-0. Epub 2014 Aug 17. PMID 25127644
- [Background] Buitelaar J, Bolte S, Brandeis D, Caye A, Christmann N, Cortese S, Coghill D, Faraone SV, Franke B, Gleitz M, Greven CU, Kooij S, Leffa DT, Rommelse N, Newcorn JH, Polanczyk GV, Rohde LA, Simonoff E, Stein M, Vitiello B, Yazgan Y, Roesler M, Doepfner M, Banaschewski T. Toward Precision Medicine in ADHD. Front Behav Neurosci. 2022 Jul 6;16:900981. doi: 10.3389/fnbeh.2022.900981. eCollection 2022. PMID 35874653